CLINICAL TRIAL: NCT00931463
Title: A Randomised Open-label Study Comparing the Safety and Efficacy of Ritonavir Boosted Lopinavir and 2-3N(t)RTI Backbone Versus Ritonavir Boosted Lopinavir and Raltegravir in Participants Virologically Failing First-line NNRTI/2N(t)RTI Therapy
Brief Title: A Trial of 2 Options for Second Line Combination Antiretroviral Therapy Following Virological Failure of a Standard Non-nucleoside Reverse Transcriptase Inhibitor (NNRTI)+2N(t)RTI First Line Regimen
Acronym: SECOND-LINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kirby Institute (Other Government)
Collaborators: Merck Sharp & Dohme LLC (Industry); Abbott (Industry); amfAR, The Foundation for AIDS Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SECOND-LINE
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: HIV Infections
Keywords: second line therapy; combination antiretroviral therapy; first-line failure; AIDS; treatment experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Raltegravir Potassium; Nucleosides; Nucleotides; lopinavir-ritonavir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ritonavir-boosted lopinavir and 2N(t)RTI (Active Comparator): This is the current standard of care for second line therapy following failure of standard first-line NNRTI+2N(t)RTIs according to WHO guidelines.
  Interventions: Drug: 2N(t)RTI; Drug: Ritonavir-boosted lopinavir
- Ritonavir-boosted lopinavir and raltegravir (Experimental): This is an experimental arm which is likely to be fully active in the presence of N(t)RTI mutations and which preliminary evidence suggests should be potent and durable.
  Interventions: Drug: raltegravir; Drug: Ritonavir-boosted lopinavir

INTERVENTIONS:
Drug: raltegravir — 400 mg raltegravir tablet taken every 12 hours
  Other Names: Isentress
  Arms: Ritonavir-boosted lopinavir and raltegravir
Drug: 2N(t)RTI — 2N(t)RTIs as prescribed
  Other Names: nucleosides, nucleotides, nuncleoside backbone
  Arms: Ritonavir-boosted lopinavir and 2N(t)RTI
Drug: Ritonavir-boosted lopinavir — 2 heat-stable tablets of ritonavir-boosted lopinavir taken every 12 hours
  Other Names: Aluvia, Kaletra

SUMMARY:
The investigators hypothesize that following virological failure of a standard NNRTI+2N(T)RTI regimen second-line antiretroviral therapy consisting of ritonavir-boosted lopinavir and 2N(T)RTIs will offer comparable efficacy to that provided by ritonavir-boosted lopinavir and raltegravir.

The study will be conducted for 96-weeks with the primary endpoint analyzed after 48-weeks.

The primary endpoint is virological: a comparison of virological suppression in plasma < 200 copies/mL between the randomized arms after 48 weeks.

Secondary and exploratory endpoints include virological, immunological, safety, clinical, metabolic, drug adherence, drug resistance and quality of life.

DETAILED DESCRIPTION:
In HIV-infected subjects who have virologically failed first-line antiretroviral therapy comprising 2N(t)RTI + NNRTI a regimen of second-line therapy incorporating ritonavir-boosted lopinavir and raltegravir provides comparable (i.e., non-inferior) antiretroviral efficacy over 48 weeks to a regimen containing ritonavir-boosted lopinavir and 2-3N(t)RTIs.

Eligible patients will be randomised to one of two arms:

I. ritonavir boosted lopinavir (LPV/r) 200mg/50mg 4 tabs once daily or 2 tabs twice daily + 2-3N(t)RTIs

II. ritonavir boosted lopinavir (LPV/r) 200mg/50mg 4 tabs once daily or 2 tabs twice daily + raltegravir 400 mg twice daily

The primary objective of this study is to compare the virological efficacy of the two strategies as measured by the proportion of participants with HIV RNA < 200 copies/mL 48 weeks after randomisation.

Secondary objectives include virological, immunological, safety and antiretroviral therapy endpoints.

Exploratory endpoints include clinical, metabolic, drug resistance, medication adherence and quality of life endpoints.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-1 positive by licensed diagnostic test
2. Aged 16 years or older (or minimum age as determined by local regulations or as legal requirements dictate)
3. Have received first antiretroviral regimen consisting of an NNRTI plus 2N(t)RTIs for at least 24 weeks
4. No change in antiretroviral therapy within 12 weeks prior to screening
5. Failed first-line NNRTI + 2N(t)RTI combination therapy according to virological criteria defined by two consecutive (at least 7 days apart) HIV RNA results of greater then 500 copies/mL
6. No prior or current exposure to HIV protease inhibitors and/or HIV integrase inhibitors
7. Able to provide written informed consent

Exclusion Criteria:

1. The following laboratory variables:

   * absolute neutrophil count (ANC) < 500 cells/microlitres
   * hemoglobin < 7.0 g/decilitres
   * platelet count < 50,000 cells/microlitres
   * ALT great than 5 x ULN
2. Pregnant or nursing mothers
3. Participants with active viral hepatitis B infection defined by the presence in serum of hepatitis B surface antigen
4. Use of immunomodulators within 30 days prior to screening
5. Use of any prohibited medications (rifampicin, midazolam, triazolam, cisapride, pimozide, amiodarone, dihydroergotamine, ergotamine, ergonovine, methylergonovine, astemizole, terfenadine, vardenafil, and St. John's wort)
6. Intercurrent illness requiring hospitalization
7. Active opportunistic disease not under adequate control in the opinion of the site Principal Investigator
8. Participants with current alcohol or illicit substance abuse that in the opinion of the site Principal Investigator might adversely affect participation in the study
9. Participants deemed by the site Principal Investigator unlikely to be able to remain in follow-up for the protocol-defined period

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 558 (Actual)
Dates: Start 2009-09; Primary Completion 2012-09 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Cooper, MD, Study Chair — Kirby Institute; Brian Gazzard, MD, Study Chair — St. Stephen's Trust
Locations (44):
- Argentina (10):
  - Hospital Interzonal General de Agudos, Oscar Alende, Buenos Aires, Mar Del Plata Provincia
  - CAICI, Buenos Aires, Rosario Provincia de Sante Fe
  - Hospital General de Agudos 'Teodoro Alvarez', Buenos Aires
  - FUNCEI, Buenos Aires
  - Hospital de Infecciosas FJ Muniz, Buenos Aires
  - Hospital Italiano, Buenos Aires
  - Hospital J.M. Ramos Mejia, Buenos Aires
  - Hospital Prof. Alejandro Posadas, Buenos Aires
  - Hospital Rawson, Córdoba
  - Hospital Central, Mendoza
- Australia (5):
  - Liverpool Hospital, Liverpool, New South Wales
  - Albion Street Centre, Sydney, New South Wales
  - St Vincent's Hospital, Sydney, New South Wales
  - The Alfred Hospital, Melbourne, Victoria
  - Centre Clinic, Melbourne, Victoria
- Chile (2):
  - Hospital de la Universidad Catolica Pontificia, Santiago
  - Hospital San Borja-Arriaran, Santiago
- Hopital Saint-Louis, Paris, France
- Germany (2):
  - Medical Group Practice, Berlin
  - J W Goethe Universitat, Frankfurt
- Queen Elizabeth Hospital, Hong Kong, Kowloon, Hong Kong
- India (2):
  - YRG Care, Chennai
  - Institute of Infectious Diseases, Pune
- Mater Misericordiae-Dublin, Dublin, Ireland
- Malaysia (3):
  - Hospital Pelau Pinang, Kuala Lumpur
  - Hospital Sungai Buloh, Kuala Lumpur
  - University of Malaysia, Kuala Lumpur
- Mexico (3):
  - Hospital General de Guadalajara, Guadalajara
  - Hospital General de Leon, León
  - Instituto Nacional de Ciencias Medicas y Nutricion "Salvado Zubiran", Mexico City
- Auckland Hospital, Grafton, Auckland, New Zealand
- Nigeria (3):
  - Evangel Hospital (ECWA), Jos, Plateau State
  - Jos University Teaching Hospital (JUTH), Jos, Plateau State
  - Plateau State Specialist Hospital, Jos, Plateau State
- Peru (4):
  - Hospital Almenara, Lima
  - IMPACTA/Hospital Dos de Mayo, Lima
  - Instituto de Medicina Tropical Alexander von Humboldt, Universidad Peruana Cayetano Heredia, Lima
  - Via Libre, Lima
- Tan Tock Seng Hospital, Singapore, Singapore
- South Africa (3):
  - Josha Research, Bloemfontein
  - Desmond Tutu HIV Foundation, Cape Town
  - Chris Hani Baragwanath Hospital, Soweto
- National Taiwan University Hospital, Taipei, Taiwan
- Chelsea and Westminster Hospital, Fulham, London, United Kingdom

REFERENCES:
- [Derived] Henry RT, Jiamsakul A, Law M, Losso M, Kamarulzaman A, Phanuphak P, Kumarasamy N, Foulkes S, Mohapi L, Nwizu C, Wood R, Kelleher A, Polizzotto M; SECOND-LINE Study Group. Factors Associated With and Characteristic of HIV/Tuberculosis Co-Infection: A Retrospective Analysis of SECOND-LINE Clinical Trial Participants. J Acquir Immune Defic Syndr. 2021 May 1;87(1):720-729. doi: 10.1097/QAI.0000000000002619. PMID 33399309
- [Derived] Amin J, Boyd MA, Kumarasamy N, Moore CL, Losso MH, Nwizu CA, Mohapi L, Kerr SJ, Sohn AH, Teppler H, Renjifo B, Molina JM, Emery S, Cooper DA. Raltegravir non-inferior to nucleoside based regimens in second-line therapy with lopinavir/ritonavir over 96 weeks: a randomised open label study for the treatment of HIV-1 infection. PLoS One. 2015 Feb 27;10(2):e0118228. doi: 10.1371/journal.pone.0118228. eCollection 2015. PMID 25723472
- [Derived] Martin A, Moore CL, Mallon PW, Hoy JF, Emery S, Belloso WH, Phanuphak P, Ferret S, Cooper DA, Boyd MA; Second-Line Study Team. HIV lipodystrophy in participants randomised to lopinavir/ritonavir (LPV/r) +2-3 nucleoside/nucleotide reverse transcriptase inhibitors (N(t)RTI) or LPV/r + raltegravir as second-line antiretroviral therapy. PLoS One. 2013 Oct 30;8(10):e77138. doi: 10.1371/journal.pone.0077138. eCollection 2013. PMID 24204757
- [Derived] SECOND-LINE Study Group; Boyd MA, Kumarasamy N, Moore CL, Nwizu C, Losso MH, Mohapi L, Martin A, Kerr S, Sohn AH, Teppler H, Van de Steen O, Molina JM, Emery S, Cooper DA. Ritonavir-boosted lopinavir plus nucleoside or nucleotide reverse transcriptase inhibitors versus ritonavir-boosted lopinavir plus raltegravir for treatment of HIV-1 infection in adults with virological failure of a standard first-line ART regimen (SECOND-LINE): a randomised, open-label, non-inferiority study. Lancet. 2013 Jun 15;381(9883):2091-9. doi: 10.1016/S0140-6736(13)61164-2. PMID 23769235

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place from Mar-2010 till Sept-2011 at 37 sites in Argentina, Australia, Chile, UK, France, Hong Kong, India, Israel, Malaysia, Mexico, Peru, Nigeria, Singapore, South Africa, and Thailand. The sites had to be clinical facilities with a cohort of suitable patients and able to do protocol-mandated procedures.
Pre-assignment Details: 558 participants were enrolled in the study. 14 were excluded because of unverifiable data at one site and 3 dropped out before analysis, never received study treatment
Period: Overall Study
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Started | 271 | 270
Completed | 254 | 265
Not Completed | 17 | 5
Not completed — Death | 8 | 4
Not completed — Withdrawal by Subject | 5 | 0
Not completed — Lost to Follow-up | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Ritonavir-boosted Lopinavir and 2N(t)RTI: Lopinavir / ritonavir + 2-3N(t)RTI: LPV/r 200mg/50mg 4 tabs once daily or 2 tabs twice daily + 2-3 N(t)RTI
- Ritonavir-boosted Lopinavir and Raltegravir: Lopinavir /ritonavir + raltegravir: LPV/r 200mg/50mg 4 tabs once daily or 2 tabs twice daily + raltegravir 400mg 1 tablet twice daily
- Total: Total of all reporting groups
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir | Total
Number analyzed (Participants) | 271 | 270 | 541
Age, Continuous [Mean (Standard Deviation); unit: years] | 39 (8.81) | 38.55 (8.84) | 38.78 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 128 | 243
  Male | 156 | 142 | 298
Region of Enrollment [Number; unit: participants]
  Africa | 100 | 96 | 196
  Southeast Asia | 116 | 113 | 229
  Europe | 1 | 2 | 3
  Australia | 1 | 0 | 1
  South America | 53 | 59 | 112

OUTCOME MEASURES:

1. Primary Outcome: Participants With Plasma HIV RNA < 200 Copies/mL 48 Weeks After Randomization
Time Frame: 48 weeks following randomization
Population: modified intention-to-treat
Measure: Number; unit: participants
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Number analyzed (Participants) | 271 | 270
participants | 219 | 223

2. Secondary Outcome: Participants With Plasma HIV RNA < 200 Copies/mL 48 Weeks After Randomization, Per-protocol Population
Description: The per- protocol population includes those participants who fulfil the protocol in the terms of the eligibility, interventions, and outcome assessment
Time Frame: 48 weeks
Population: Per protocol
Measure: Number; unit: participants
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Number analyzed (Participants) | 249 | 246
participants | 211 | 211

3. Secondary Outcome: Participants With Plasma HIV RNA < 200 Copies/mL 48 Weeks After Randomization, Per-protocol Population, Non-completer Classed as Failure
Description: The non-completer classed as failure analysis will include all randomised participants; participants who meet the following criteria will be defined as failures:
  i. week 48 HIV RNA being above each threshold ii. has missing HIV-1 RNA data for any reason iii. stops randomly assigned therapy
Time Frame: 48 weeks
Population: Non-completer classes as failure
Measure: Number; unit: participants
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Number analyzed (Participants) | 271 | 270
participants | 208 | 210

4. Secondary Outcome: Participants With Plasma HIV RNA < 200 Copies/mL 48 Weeks After Randomization, Per-protocol Population, Baseline VL >100,000 Copies Per mL
Description: The difference between treatment arms in proportion of participants with plasma HIV RNA < 200 copies/mL 48 weeks after randomization, per-protocol population: stratified analysis by baseline plasma viral load (less than or equal to 100,000 copies per mL or >100,000 copies per mL) on those participants who fulfil the protocol in the terms of the eligibility, interventions, and outcome assessment
Time Frame: 48 weeks
Population: Baseline viral load >100,000 copies per mL
Measure: Number; unit: participants
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Number analyzed (Participants) | 52 | 60
participants | 31 | 39

5. Secondary Outcome: Participants With Plasma HIV RNA < 200 Copies/mL 48 Weeks After Randomization, Per-protocol Population, VL Less Than or Equal to 100,000 Copies Per mL
Description: as for outcome 2
Time Frame: 48 weeks
Population: Baseline viral load <=100,000 copies per mL
Measure: Number; unit: participants
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Number analyzed (Participants) | 219 | 210
participants | 188 | 184

ADVERSE EVENTS:
Time Frame: 96 weeks
Description: AEs reported by investigators
Arm/Group | Ritonavir-boosted Lopinavir and 2N(t)RTI | Ritonavir-boosted Lopinavir and Raltegravir
Serious Adverse Events (participants affected / at risk) | 23/271 | 24/270
Other Adverse Events (participants affected / at risk) | 243/271 | 232/270
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ritonavir-boosted Lopinavir and 2N(t)RTI (N=271) | Ritonavir-boosted Lopinavir and Raltegravir (N=270)
Acute gastroenteritis (Gastrointestinal disorders) | 0 | 2
Abdominal Pain- death (Gastrointestinal disorders) | 1 | 0
Acute Asthma Attack (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Asymptomatic neuro-syphillis (Nervous system disorders) | 1 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CIN II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
CMV Retinitis (Infections and infestations) | 1 | 1
Car accident - resulted in death (Injury, poisoning and procedural complications) | 0 | 1
Contusions resulting in hospitalisations (Injury, poisoning and procedural complications) | 0 | 1
Cervical cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Convulsions (General disorders) | 0 | 1
Cryptococcal meningitis (Infections and infestations) | 0 | 1
Cryptococcal disseminated (Infections and infestations) | 1 | 0
Death - unknown, possible due to recurrent anaemia, HIV disease (Blood and lymphatic system disorders) | 0 | 1
Death, cause unknown (General disorders) | 2 | 1
Death, probably due to myocardial infarction (General disorders) | 0 | 1
Delirium, secondary alcohol withdrawal (Social circumstances) | 0 | 1
Dysentery (Gastrointestinal disorders) | 1 | 0
Extrapulmonary TB - resulted in death (Infections and infestations) | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0
Fracture of right ankle (Injury, poisoning and procedural complications) | 0 | 1
Gangrenous bowel (Gastrointestinal disorders) | 1 | 0
Giardiasis and nocardiasis resulting in death (Infections and infestations) | 1 | 0
HSV meningitis (Infections and infestations) | 0 | 1
herpez zoster (Infections and infestations) | 0 | 1
haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Varizella zoster infection and MSSA cervical lymphadenitis (Infections and infestations) | 1 | 0
Fever and anaemia hospitalization (Blood and lymphatic system disorders) | 1 | 0
Haematoma inside lower colon (Blood and lymphatic system disorders) | 1 | 0
Skin graft detachment (Surgical and medical procedures) | 0 | 1
hyponatremia (Metabolism and nutrition disorders) | 1 | 0
kaposi sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung abscess resulted in death (Respiratory, thoracic and mediastinal disorders) | 0 | 1
meningitis (Nervous system disorders) | 0 | 1
miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Plasmodiasis (Infections and infestations) | 1 | 0
pneumonia (Infections and infestations) | 3 | 3
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 5 | 7
Probable righ ovarian carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Genital bleeding (Reproductive system and breast disorders) | 0 | 1
Pulmonary tuberculosis (Infections and infestations) | 0 | 2
Pyelonephritis (Renal and urinary disorders) | 0 | 1
Renal failure resulted in death (Renal and urinary disorders) | 2 | 0
Right middle lobe pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sepsis (Infections and infestations) | 0 | 1
Skin ulcers superinfected (Infections and infestations) | 0 | 1
Squamous cell carcinoma of the anal canal - resulted in death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Stroke (Vascular disorders) | 0 | 1
Supra Condylar fracture of right femur (Injury, poisoning and procedural complications) | 1 | 0
Urinary tract infection (Renal and urinary disorders) | 0 | 1
TB meningitis (Infections and infestations) | 0 | 1
Tension Headache (General disorders) | 0 | 1
Uveitis (Eye disorders) | 1 | 0
Varizella zoster (Infections and infestations) | 1 | 0
Viral infection (presumptive) (Infections and infestations) | 0 | 1
Acute abdomen (Gastrointestinal disorders) | 0 | 1
Acute renal impairment (Renal and urinary disorders) | 1 | 0
Cerebral toxoplasmosis (Infections and infestations) | 0 | 1
Crytococcal meningitis and giardiasis (Infections and infestations) | 1 | 0
Diarrhoea for over consumption of alcohol (Gastrointestinal disorders) | 0 | 1
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Hemoptysis, resulted in death (Blood and lymphatic system disorders) | 0 | 1
Right side pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Bloody diarrhoea (Gastrointestinal disorders) | 1 | 0
diarrhoea (Gastrointestinal disorders) | 1 | 0
Infective diarrhoea (Infections and infestations) | 1 | 0
miliary tuberculosis (Infections and infestations) | 0 | 1
Perianal HSV ulcer (Infections and infestations) | 1 | 0
pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 0
probable PCP and presumptive mycobacterium TB (Infections and infestations) | 0 | 1
Salmonella and PCP (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ritonavir-boosted Lopinavir and 2N(t)RTI (N=271) | Ritonavir-boosted Lopinavir and Raltegravir (N=270)
Allergic conditions (General disorders) | 12 (15) | 8 (8)
Anaemias nonhaemolytic and marrow depression (Blood and lymphatic system disorders) | 10 (21) | 11 (12)
Appetite and general nutritional disorders (Metabolism and nutrition disorders) | 25 (33) | 12 (16)
Bacterial infectious disorders (Infections and infestations) | 9 (11) | 7 (7)
Body temperature conditions (General disorders) | 26 (32) | 23 (26)
Bone, calcium, magnesium and phosphorus metabolism disorders (Metabolism and nutrition disorders) | 7 (7) | 6 (6)
Decreased and nonspecific blood pressure disorders and shock (Blood and lymphatic system disorders) | 13 (13) | 15 (17)
Dental and gingival conditions (General disorders) | 2 (3) | 7 (7)
Epidermal and dermal conditions (Skin and subcutaneous tissue disorders) | 66 (108) | 66 (115)
Female reproductive tract infections and inflammations (Reproductive system and breast disorders) | 14 (18) | 15 (22)
Fungal infectious disorders (Infections and infestations) | 33 (39) | 47 (54)
Gastrointestinal inflammatory conditions (Gastrointestinal disorders) | 3 (3) | 8 (8)
Gastrointestinal motility and defaecation conditions (Gastrointestinal disorders) | 128 (177) | 102 (131)
Gastrointestinal signs and symptoms (Gastrointestinal disorders) | 72 (145) | 51 (82)
General system disorders NEC (General disorders) | 34 (47) | 33 (41)
Headaches (General disorders) | 41 (52) | 30 (36)
Hepatic and hepatobiliary disorders (Hepatobiliary disorders) | 2 (2) | 8 (8)
Infections - pathogen class unspecified (Infections and infestations) | 103 (188) | 124 (243)
Injuries NEC (Injury, poisoning and procedural complications) | 8 (8) | 13 (13)
Joint disorders (Musculoskeletal and connective tissue disorders) | 13 (15) | 22 (23)
Lipid metabolism disorders (Endocrine disorders) | 6 (6) | 7 (8)
Menstrual cycle and uterine bleeding disorders (Reproductive system and breast disorders) | 7 (8) | 11 (12)
Muscle disorders (Musculoskeletal and connective tissue disorders) | 16 (18) | 19 (23)
Musculoskeletal and connective tissue disorders NEC (Musculoskeletal and connective tissue disorders) | 39 (51) | 44 (53)
Neurological disorders NEC (Nervous system disorders) | 10 (13) | 9 (9)
Ocular infections, irritations and inflammations (Eye disorders) | 9 (10) | 17 (22)
Oral soft tissue conditions (Skin and subcutaneous tissue disorders) | 8 (9) | 10 (11)
Pregnancy, labour, delivery and postpartum conditions (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 6 (7)
Protozoal infectious disorders (Infections and infestations) | 21 (40) | 13 (30)
Renal disorders (excl nephropathies) (Renal and urinary disorders) | 8 (9) | 2 (3)
Reproductive tract disorders NEC (Reproductive system and breast disorders) | 4 (4) | 12 (12)
Respiratory disorders NEC (Respiratory, thoracic and mediastinal disorders) | 51 (77) | 58 (112)
Skin appendage conditions (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (9)
Sleep disorders and disturbances (General disorders) | 12 (12) | 8 (8)
Vascular haemorrhagic disorders (Vascular disorders) | 12 (13) | 9 (10)
Vascular hypertensive disorders (Vascular disorders) | 4 (4) | 11 (11)
Viral infectious disorders (Infections and infestations) | 40 (53) | 41 (56)
Vulvovaginal disorders (excl infections and inflammations) (Reproductive system and breast disorders) | 7 (9) | 8 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is a Clinical Trial Agreement signed with each PI detailing the publication policy and disclosure of study's information, in summary:

* The Institution, its personnel and the Principal Investigator must not Publish or present any aspect of the Study without the prior written approval of the sponsor, except for the purposes of internal training
* Publications or presentations of results from the Study will follow the agreement's publication/presentation guidelines